CLINICAL TRIAL: NCT06760819
Title: A Phase 2 Open-label Basket Study to Evaluate the Efficacy and Safety of Orally Administered Reversible Tyrosine Kinase Inhibitor BAY 2927088 in Participants With Metastatic or Unresectable Solid Tumors With HER2-activating Mutations
Brief Title: A Study to Learn More About How Well Treatment With Sevabertinib (BAY 2927088) Tablets Works and How Safe it is in Participants Who Have a Solid Tumor With Mutations of the Human Epidermal Growth Factor Receptor 2 (HER2)
Acronym: panSOHO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22752; 2024-517419-62-00 (Registry Identifier: CTIS (EU))
Expanded Access: NCT06761976 (Available)
Record Dates: First submitted 2024-12-18; First posted 2025-01-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors; HER2 Mutation
Keywords: Colorectal cancer; CRC; Biliary tract cancer; BTC; Bladder cancer; Cervical cancer; Endometrial cancer; Sarcoma; Gastrointestinal stromal tumor; GIST; Breast cancer; Gastrointestinal cancer; GI cancer; Gastric cancer; Esophageal cancer; Gallbladder cancer; Pancreatic cancer; Ovarian Cancer; Salivary cancer; Ampullary cancer; Urothelial cancer; HER2 mutant cancer
MeSH Terms: conditions — Colorectal Neoplasms; Biliary Tract Neoplasms; Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Sarcoma; Gastrointestinal Stromal Tumors; Breast Neoplasms; Gastrointestinal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Gallbladder Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY2927088 (Experimental): Adult participants with metastatic or unresectable solid tumors with HER-2 activating mutations including: colorectal, biliary tract, bladder, cervical, endometrial, breast, and other solid tumor types. Participants will receive BAY2927088 20 mg BID until disease progression per RECICST 1.1, unacceptable toxicity, or until any other withdrawal criteria.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BID: twice a day
  Interventions: Drug: BAY2927088

INTERVENTIONS:
Drug: BAY2927088 — tablet, oral
  Other Names: Sevabertinib

SUMMARY:
Researchers are looking for a better way to treat people who have solid tumors with HER2-activating mutations. Before a treatment can be approved for people to take, researchers do clinical trials to better understand its safety and how it works.

In this trial, the researchers want to learn how well BAY2927088 (sevabertinib) works in people with different types of solid tumors with HER2 mutations. These include tumors in the colon or rectum, the uterus and the cervix (lower part of the uterus), the breast, the bladder, and the biliary tract (includes gall bladder and bile ducts) as well as other types of solid tumors with the exception of people with advanced non-small cell lung cancer (NSCLC).

Solid tumors may have specific changes or mutations to a gene called human epidermal growth receptor-2 (HER2). This leads to the formation of an abnormal form of HER2 protein in the cancer cells, resulting in increased cell growth. The study treatment, BAY2927088, is expected to block the abnormal HER2 protein which may stop the spread of cancer.

The trial will include about 111 participants who are at least 18 years old. All the participants will take 20 mg of BAY2927088 as tablets by mouth.

The participants will take treatments in 3-week periods called cycles. These 3-week cycles will be repeated throughout the trial. The participants can take BAY2927088 until their cancer gets worse, until they have medical problems, or until they leave the trial.

During the trial, the doctors will take imaging scans of different parts of the body to study the spread of cancer and will check heart health using echocardiogram or cardiac magnetic resonance imaging (MRI) and electrocardiogram (ECG). The doctors will also take blood and urine samples and do physical examinations to check the participants' health. They will ask questions about how the participants are feeling and if they have any medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically or cytologically confirmed locally advanced, unresectable or metastatic solid tumor cancer (colorectal carcinoma; biliary tract cancer; bladder and urothelial tract cancer; cervical cancer; endometrial cancer; breast cancer; other solid tumor cancer, excluding NSCLC)
* Participant must be ≥18 years of age or over the legal age of consent
* Patients who have received prior standard therapy appropriate for their tumor type and stage of disease, or who have no satisfactory alternative treatments
* Documented activating HER2 mutation
* At least one measurable lesion that would qualify as a target lesion by RECIST 1.1 criteria

Exclusion Criteria:

* Primary diagnosis of non-small cell lung cancer (NSCLC)
* Prior treatment with a HER2 tyrosine kinase inhibitor (TKI)
* Active brain metastases
* Uncontrolled, severe, intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 as assessed by BICR | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  ORR is defined as the proportion of participants with a best overall response of confirmed complete response (CR) or partial response (PR) per RECIST 1.1 by BICR. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have decreased in size to have a short axis of <10 mm. PR is defined as a ≥30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BICR = blinded independent central review (BICR)

SECONDARY OUTCOMES:
Duration of response (DOR) per RECIST 1.1 as assessed by BICR | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  DOR is defined as the time from date of first documented complete or partial response (if confirmed) until the earliest date of progressive disease (PD) per RECIST 1.1 as assessed by BICR, or death from any cause, whichever occurs first. PD is defined as a ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BICR = blinded independent central review (BICR)
Time to response (TTR) per RECIST 1.1 as assessed by BICR | From first participant enrolled until end of treatment or end of imaging active follow-up (up to approximately 3 years)
  TTR is defined as the time from the start of study treatment until the date of first documented complete or partial response (if confirmed) per RECIST 1.1 as assessed by BICR.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BICR = blinded independent central review (BICR)
ORR per RECIST 1.1 as assessed by the investigator | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  ORR is defined as the proportion of participants with a best overall response of confirmed CR or confirmed PR per RECIST 1.1 by investigator.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1
Disease control rate (DCR) per RECIST 1.1 as assessed by BICR | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  DCR is defined as the proportion of participants with a best overall response of confirmed complete response (CR) or partial response (PR) or stable disease (SD), by the BICR per RECIST 1.1. SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
DCR ≥12 weeks per RECIST 1.1 as assessed by BICR | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  Defined as the proportion of participants with a best overall response of confirmed CR or PR or SD (for at least 12 weeks following the first study intervention), by the BICR per RECIST 1.1.
Progression-free survival (PFS) per RECIST 1.1 as assessed by BICR | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  Defined as the time from date of start of treatment until the earliest date of PD per RECIST 1.1 as assessed by the BICR, or death from any cause, whichever occurs first.
Disease control rate (DCR) per RECIST 1.1 as assessed by the investigator | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  Defined as the proportion of participants with a best overall response of confirmed CR or PR or SD, by the investigator per RECIST 1.1.
DCR ≥12 weeks per RECIST 1.1 as assessed by the investigator | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  Defined as the proportion of participants with a best overall response of confirmed CR or PR or SD (for at least 12 weeks following the first study intervention), by the investigator per RECIST 1.1.
Progression-free survival (PFS) per RECIST 1.1 as assessed by the investigator | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  Defined as the time from date of start of treatment until the earliest date of PD per RECIST 1.1 as assessed by the investigator, or death from any cause, whichever occurs first
DOR per RECIST 1.1 as assessed by the investigator | From start of study intervention until the first documented progression, or death from any cause, or end of study (up to approximately 3 years), whichever comes first
  DOR is defined as the time from date of first documented complete or partial response (if confirmed) until the earliest date of PD per RECIST 1.1 as assessed by the investigator, or death from any cause, whichever occurs first.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1
TTR per RECIST 1.1 as assessed by the investigator | From first participant enrolled until end of treatment or end of imaging active follow-up (up to approximately 3 years)
  TTR is defined as the time from the start of study treatment until the date of first documented complete or partial response (if confirmed) per RECIST 1.1 as assessed by the investigator.
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1
Overall survival (OS) | From start of study intervention until death from any cause, or end of study (up to approximately 3 years), whichever comes first
  Defined as the time from the start of study treatment to the date of death from any cause.
Number of participants with treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) per CTCAE v 5.0, categorized by severity, including number of participants who discontinue study treatment due to an AE | From first participant enrolled until up to 30 days after the last administration of study treatment
  From first administration of study intervention up to 30 days after the last dose of study intervention.
Time to deterioration in EORTC QLQ-C30 physical functioning domain score | Baseline and up until end of treatment or end of imaging active follow-up (up to approximately 3 years)
  The EORTC QLQ-C30 is a multi-dimensional validated cancer-specific quality of life (QoL) questionnaire developed by the EORTC Study Group on QoL for use in international clinical trial settings. The EORTC QLQ-C30 will be used to evaluate the time to deterioration in the physical functioning domain score.
  EORTC QLQ-C30 = European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30
Change from baseline in EORTC QLQ-C30 physical functioning domain score | Baseline and up until end of treatment or end of imaging active follow-up (up to approximately 3 years)
  The EORTC QLQ-C30 is a multi-dimensional validated cancer-specific quality of life (QoL) questionnaire developed by the EORTC Study Group on QoL for use in international clinical trial settings. The EORTC QLQ-C30 will be used to evaluate the change from baseline in the physical functioning domain score.
  EORTC QLQ-C30 = European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30
Change from baseline in EORTC QLQ-C30 global health status/quality of life (QoL) | Baseline and up until end of treatment or end of imaging active follow-up (up to approximately 3 years)
  The EORTC QLQ-C30 is a multi-dimensional validated cancer-specific quality of life (QoL) questionnaire developed by the EORTC Study Group on QoL for use in international clinical trial settings. The EORTC QLQ-C30 will be used to evaluate the change from baseline in global health status/QoL.
  EORTC QLQ-C30 = European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30

CONTACTS AND LOCATIONS:
Locations (54):
- United States (11):
  - UAB O'Neal Comprehensive Cancer Center - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - City of Hope - Duarte Cancer Center, Duarte, California
  - Florida Cancer Specialists & Research Institute - Fort Myers Cancer Center - Gladiolus, Fort Myers, Florida
  - Dana-Farber Cancer Institute - Oncology Department, Boston, Massachusetts
  - Brigette Harris Cancer Pavilion at Henry Ford Cancer Center - Detroit, Detroit, Michigan
  - Profound Research -OMG - TriAtria Cancer Center, Farmington Hills, Michigan
  - Cleveland Clinic - Oncology Department, Cleveland, Ohio
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - Gynecology Oncology clinic at UW Medical Center - Montlake, Seattle, Washington
  - UW Health Carbone Cancer Center, Madison, Wisconsin
- Australia (3):
  - NSW Health - Blacktown Hospital, Blacktown, New South Wales
  - Macquarie University Hospital - Oncology Department, Sydney, New South Wales
  - ICON Cancer Centre - Southport, Southport, Queensland
- Canada (3):
  - Queen Elizabeth II Health Sciences Centre - Victoria General Site, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre - University Health Network - Department of Medical Oncology and Hematology, Toronto, Ontario
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- China (6):
  - Peking University First Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Cancer Hospital - Oncology Department, Beijing, Beijing Municipality
  - Hunan Cancer Hospital - Oncology Department, Changsha, Hunan
  - Zhongshan Hospital, Fudan University - Oncology Department, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang Univ. School of Medicine - Oncology Department, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center - Oncology Department, Shanghai
- Denmark (3):
  - Aarhus University Hospital - Oncology Department, Aarhus N
  - Rigshospitalet - Kræftbehandling, Copenhagen
  - Odense University Hospital - Oncology Department, Odense C
- France (6):
  - Institut Bergonie - Unicancer Nouvelle Aquitaine - Service Oncologie medicale, Bordeaux
  - CHU Brest - Hopital La Cavale Blanche - service oncologie medicale, Brest
  - Centre Oscar Lambret - Service Oncologie, Lille
  - ICM - Institut du Cancer de Montpellier - Val d'Aurelle - CIPP, Montpellier
  - Centre Hospitalier Lyon Sud - Service oncologie medicale, Pierre-Bénite
  - Institut Gustave Roussy - Departement d'Innovation Therapeutique et d'Essais Precoces (DITEP), Villejuif
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S. C. Oncologia Medica 1, Milan
  - Istituto Europeo di Oncologia s.r.l - Ginecologia Oncologica Medica, Milan
  - Azienda USL IRCCS di Reggio Emilia_Arcispedale Santa Maria Nuova - S.C. Oncologia Provinciale, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Roma
- Japan (6):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East (NCCHE) - Kashiwa Campus, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kindai University Hospital, Sakai, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- South Korea (4):
  - Severance Hospital, Yonsei University Health System - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center | Oncology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center - Oncology Department, Seoul
- Spain (5):
  - Institut Catala D'oncologia | Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad De Navarra | Oncologia Medica, Madrid, Navarre
  - Hospital Universitari Dexeus Grupo Quironsalud | Oncologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia Medica, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz | Oncologia Medica, Madrid
- Switzerland (3):
  - Inselspital Bern - Universitätsklinik für Medizinische Onkologie, Bern
  - Hopitaux Universitaires de Geneve - Oncology Department, Geneva
  - Univestitätsspital Zürich (USZ), Zurich

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.